CLINICAL TRIAL: NCT04934605
Title: A Genotype-phenotype Correlation of SLC26A4 Mutations in Cochlear-implanted Patients With Enlarged Vestibular Aqueduct
Brief Title: Genotype-phenotype Correlation of SLC26A4 in CI Patients With EVA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-007
Record Dates: First submitted 2021-06-10; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-04

CONDITIONS: Sensorineural Hearing Loss; Enlarged Vestibular Aqueduct
Keywords: enlarged vestibular aqueduct; SLC26A4; cochlear implant
MeSH Terms: conditions — Hearing Loss, Sensorineural; Deafness, Autosomal Recessive 4 | interventions — Cochlear Implantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cochlear implantation — Cochlear implantation

SUMMARY:
To explore the genotype-phenotype correlation of SLC26A4 mutations in cochlear-implanted patients with enlarged vestibular aqueduct.

DETAILED DESCRIPTION:
Enlarged vestibular aqueduct (EVA) is one of the most common forms of inner ear malformation that cause sensorineural hearing loss (SNHL). Some patients with EVA present delayed, fluctuating, and progressive hearing loss, while the others are with congenital or sudden hearing loss. Cochlear implants (CI) have been widely used in patients with severe-profound SNHL. However, it is difficult to define the optimal timing of CI operations for patients with EVA. Mutations in SLC26A4 are known to be responsible for EVA. This study is to explore the genotype-phenotype correlation of SLC26A4 mutations in cochlear-implanted patients with EVA.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral severe-to-profound sensorineural hearing loss who received cochlear implantation.
2. Bilateral or unilateral enlarged vestibular aqueduct (EVA) with or without Mondini malformation (IP-II) on temporal bone computed tomography (CT) and/or magnetic resonance imaging (MRI).

Exclusion Criteria:

1. Hearing loss that is associated with symptoms which meet the criteria of already known syndromes.
2. With other type of inner ear malformation.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with sensorineural hearing loss and enlarged vestibular aqueduct.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Cochlear implant age | Immediately after cochlear implantation
  Age of cochlear implantation.
Duration of hearing loss | Immediately after cochlear implantation
  Time between found of hearing loss and cochlear implantation.

SECONDARY OUTCOMES:
Type of initial hearing loss | On the 1 day of recruitment.
  Prelingual or postlingual; Hearing aid can or cannot benefit
Type of hearing loss progression | Immediately after cochlear implantation
  Initial profound, sudden, or fluctuating hearing loss.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Liu, MD, Principal Investigator — Department of Otorhinolaryngology, 2nd Affiliated Hospital, School of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: Undecided